CLINICAL TRIAL: NCT06171659
Title: FDG PET/MR Imaging of Peripheral Pain Generators in Persistent Post-Surgical Pain (PPSP)
Brief Title: FDG PET/MR Imaging of Peripheral Pain Generators
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Arthroscopy Association of North America (AANA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-0884; R01AR077706 (NIH); SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison); Protocol Version 11/1/2024 (Other: UW Madison)
Record Dates: First submitted 2023-12-04; First posted 2023-12-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Pain; Nociceptive Pain
MeSH Terms: conditions — Pain; Nociceptive Pain | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Open Surgical Procedure (Arthroplasty): PPSP subjects who have undergone hip (or knee) joint arthroplasty (i.e., open surgical procedure for joint replacement).
  * 6 month post-op scans
  * 12 month post-op scans
  * 18 month post-op scans
  Interventions: Drug: FDG radiotracer; Device: PET/MRI; Device: PET/CT imaging
- Less Invasive Procedure (Arthroscopy): PPSP subjects who have undergone hip (or knee) arthroscopy (i.e., less invasive joint surgical procedure involving scopes and lower profile surgical tools)
  - 6 month post-op scans
  Interventions: Drug: FDG radiotracer; Device: PET/MRI; Device: PET/CT imaging
- Asymptomatic: Had Total Joint Replacement (Arthroplasty): Asymptomatic subjects who have undergone total hip or total knee arthroplasty.
  - single scan during one study visit (up to 3.5 hours)
  Interventions: Drug: FDG radiotracer; Device: PET/MRI; Device: PET/CT imaging
- Asymptomatic: Less Invasive Procedure (Arthroscopy): Asymptomatic subjects who have undergone hip or knee arthroscopy.
  - single scan during one study visit (up to 3.5 hours)
  Interventions: Drug: FDG radiotracer; Device: PET/MRI; Device: PET/CT imaging

INTERVENTIONS:
Drug: FDG radiotracer — Fludeoxyglucose F 18 Injection is a positron emitting radiopharmaceutical containing no-carrier added radioactive 2-deoxy-2-[18F]fluoro-D-g1ucose, which is used for diagnostic purposes in conjunction with Positron Emission Tomography (PET). It is administered by intravenous injection. Dosage planned 0.14 mCi/kg/patient.
  Other Names: fluorodeoxyglucose; 18F-Fluorodeoxyglucose
Device: PET/MRI — positron emission tomography and magnetic resonance imaging
Device: PET/CT imaging — positron emission tomography and computed tomography imaging

SUMMARY:
The purpose of this research is to determine if a PET/MRI scan using FDG can accurately identify the source of chronic pain. Identifying the source of pain may help doctors treat chronic pain more effectively. Approximately 128 participants will be enrolled and can expect to be on study for up to 12 months.

DETAILED DESCRIPTION:
The investigators aim to precisely localize sites of increased inflammation and potentially pain generation and improve understanding of nociception and inflammation using a unique, hybrid PET/MRI approach in conjunction with intravenously, administered fluorodeoxyglucose (FDG), which has been shown with PET imaging to be an sensitive surrogate marker of inflammation.

The Primary Objective of this pilot prospective, observational research is to determine whether this approach, which combines PET/MRI and an FDA-approved radiotracer, 18F-Fluorodeoxyglucose (FDG), can accurately localize the sites of painful inflammation in individuals with persistent pain.

* Determine if increased FDG uptake on PET as measured by standard uptake value (SUV) or target-to-background (TTB) measurements is increased in area of pain symptoms when compared to same corresponding areas in healthy, asymptomatic volunteers.
* Determine whether amount of FDG uptake as measured on PET is able to localize to abnormalities when compared to MR imaging (T2 signal intensity, morphologic aberrations)

Secondary Objectives:

* Verify that the standard administered adult dose of FDG (0.14 mCi/kg/patient) used currently in the clinics can also be used to detect peripheral pain generators.
* Verify that FDG uptake in asymptomatic, healthy controls will be significantly less than their chronic pain cohorts at the same anatomic location.
* Determine whether longitudinal FDG PET/MR imaging findings in individual patients directly correlate with symptoms as they evolve over time in joint arthroplasty subjects with PPSP.
* Determine if FDG PET/MR imaging findings spatially differ between different pain types.

ELIGIBILITY:
Inclusion Criteria: Persistent Post-Surgical Pain Patients

* 18-85 years old
* Presents with persistent pain with pain score of ≥4 on Numerical Rating Scale [0:10] for at least 6 months following joint arthroplasty or arthroscopy.
* Able and willing to provide informed consent
* Willing and able to undergo PET/MRI (arthroplasty and arthroscopy participants) and PET/CT (arthroplasty participants only)

Inclusion Criteria: Asymptomatic controls

* 18-85 years old
* Asymptomatic (pain score of ≤2 on the NRS) for at least 6 months following joint arthroplasty or arthroscopy.
* Able and willing to provide informed consent
* Willing and able to undergo PET/MRI

Exclusion Criteria:

* Inability to understand and communicate with the investigators to complete the study-related questionnaires.
* Any co-morbidity which results in severe systemic disease limiting function as defined by the American Society of Anesthesiology (ASA) physical status classification > 3, such as the presence of current or past (6 months) pulmonary, hepatic, renal disease, arthritis, hematopoietic, and neurological diseases not related to chronic pain.
* Pregnant or breastfeeding. (Individuals with childbearing potential will be asked to verbally confirm they are not pregnant. If they cannot confirm, they will have a urine pregnancy test either at the imaging study visit or within 7 days prior to the imaging study visit.)
* Subject with contraindication(s) to or inability to undergo PET/MRI
* Current diagnosis of malignancy of any kind. Participants in remission for at least two years and not undergoing any treatment may be considered per investigator discretion
* Current enrollment in a scientific interventional or treatment study.
* Subject unable or unwilling to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with persistent post-surgical pain and asymptomatic individuals who have undergone joint arthroplasty (hip or knee) or joint arthroscopy (hip or knee).
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in SUVmax (chronic pain) | baseline (6 months post-op), 12 months post-op, 18 months post-op
SUVmax (chronic pain vs healthy) | baseline
Location of Pain Compared to Target-to-Background (TTB) or SUVmax | baseline

SECONDARY OUTCOMES:
Number of Participants Where Standard FDG dose was sufficient to detect region of pain (symptomatic groups) | baseline
  The standard administered adult dose of FDG currently used in clinics is 0.14 mCi/kg/patient.
Variation of the maximum ratio of SUV (SUVRmax) in asymptomatic controls vs symptomatic | baseline
Variation of the maximum ratio of SUV (SUVRmax) in symptomatic participants | baseline (6 months post-op), 12 months post-op, 18 months post-op
Radiology Review Scores | up to 18 months post-op
  Radiologists will evaluate MRI and CT images from each exam, and assign 1 point to any abnormality detected in the following compartments: prosthesis itself, bone, joint space, joint capsule, muscle, subcutaneous fat, and skin, for a total of 7 possible points. Differences in scoring from MRI vs CT images will be further investigated with a t-test.
Change in Pain Scores (chronic pain) | baseline (6 months post-op), 12 months post-op, 18 months post-op
  Pain will be evaluated on a scale of 0 (no pain) to 10 (worse possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Biswal, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No